CLINICAL TRIAL: NCT03090880
Title: Long-term Prophylaxis of Venous Thromboembolism With Low-molecular-weight Heparin in Patients With Metastatic Lung Cancer
Brief Title: Prophylaxis of Venous Thromboembolism in Advanced Lung Cancer (PROVE)
Acronym: PROVE
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The rate of inclusion is too low to hope to reach the target of 800 patients. 59 patients were included, and their data will not meet the research objectives.
  The sponsor has decided to prematurely stop inclusions on January 13, 2022.
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Ministry of Health, France (Other Government); National Cancer Institute, France (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: P150963; 2016-002546-23 (EudraCT Number); PHRC (Other Grant/Funding Number: 15-059)
Record Dates: First submitted 2017-03-21; First posted 2017-03-27 (Actual); Last update posted 2022-11-17 (Actual); Status verified 2021-12

CONDITIONS: Venous Thromboembolism; Lung Neoplasm
Keywords: Low-molecular-weight Heparin; Tinzaparin
MeSH Terms: conditions — Venous Thromboembolism; Lung Neoplasms | interventions — Tinzaparin

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): usual care,
- Experimental (Experimental): tinzaparin sodium
  Interventions: Drug: Tinzaparin Sodium

INTERVENTIONS:
Drug: Tinzaparin Sodium — Subcutaneous tinzaparin 4,500 IU once daily for six months.
  Arms: Experimental

SUMMARY:
Prospective randomized open multicenter trial with blinded adjudication of endpoints to assess the efficacy of six-month low-dose LMWH (Low Molecular Weight Heparin) for the prevention of symptomatic or incidental VTE in patients with stage IV lung cancer and elevated D-dimer.

DETAILED DESCRIPTION:
Adult patients aged ≥ 18 years with stage IV lung cancer and elevated D-dimer will be randomized to the experimental or control group.Patients in the control group will receive usual care, patients in the experimental group will receive subcutaneous tinzaparin once daily for six months. Follow-up visit will take place in outpatient clinic at day 90, day 180 and day 360. Blood sampling for biomarkers will be performed at inclusion visit and day 90.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Social security affiliation
* Written informed consent
* Histologically confirmed stage IV (M1a or M1b) non-small-cell lung cancer, including recurrent non-small-cell lung cancer after a period of complete remission
* D-dimer > 1,500 µg/L
* First line of systemic cancer treatment (chemotherapy, immunotherapy or targeted therapy), or new line of systemic cancer treatment for cancer progression (chemotherapy, immunotherapy or targeted therapy), introduced during the month preceding inclusion or planned within one month after inclusion
* ECOG (Eastern Cooperative Oncology Group) score 0-2
* Life expectancy >3 months

Exclusion Criteria:

* Hypersensitivity to heparin or to any excipients
* Septic endocarditis
* History of heparin-induced thrombocytopenia
* Ongoing anticoagulant treatment at therapeutic dosage
* VTE at inclusion
* Creatinin clearance <30 mL/min
* Active bleeding
* Platelet count < 100 G/L at inclusion
* Severe hepatic insufficiency
* Cancer treated exclusively with supportive care
* Aspirin at daily dosage > 160 mg
* Pregnancy
* Patient under tutorship or curatorship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2018-09-14 (Actual); Primary Completion 2021-08-18 (Actual); Study Completion 2021-08-18 (Actual)

PRIMARY OUTCOMES:
venous thromboembolic events | 6 months
  All venous thromboembolism (VTE) events during the six-month treatment period including:
  * objectively confirmed symptomatic pulmonary embolism (PE),
  * objectively confirmed symptomatic lower-limb deep vein thrombosis (DVT) (including iliac and caval thrombosis),
  * objectively confirmed symptomatic upper extremity DVT,
  * objectively confirmed incidentally diagnosed PE or proximal DVT
  * death due to PE.

SECONDARY OUTCOMES:
Symptomatic VTE events | 6 months
  Objectively confirmed symptomatic VTE and death due to PE
Venous thromboembolic events | 12 months
  Objectively confirmed symptomatic or incidental VTE during the 12-months study period
Major bleedings | 6 months
  Major bleeding according to the ISTH criteria
Death | 6 months
  Overall mortality and causes of death
Death | 12 months
  Overall mortality and causes of death

OTHER OUTCOMES:
Risk factors for venous thromboembolism | 12 months
  Risk factors for venous thromboembolism

CONTACTS AND LOCATIONS:
Overall Officials: Guy Meyer, MD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (27):
- France (27):
  - Centre Hospitalier Annecy Genevois, Annecy, Auvergne-Rhône-Alpes
  - Hôpital Pontchaillou, Rennes, Brittany Region
  - Centre Hospitalier régional d'Orléans, Orléans, Centre-Val de Loire
  - Centre Oscar Lambret, Lille, Hauts-de-France
  - CHU de Caen, Caen, Normandy
  - CHU Poitiers, Poitiers, Nouvelle-Aquitaine
  - Hôpital Larrey, Toulouse, Occitanie
  - Institut de cancérologie de l'Ouest, Saint-Herblain, Pays de la Loire Region
  - Groupement Hospitalier Est Hospices civils de Lyon, Lyon, Rhônes Alpes
  - Institut de Cancérologie Lucien Neuwirth, Saint-Priest, Rhônes-Alpes
  - CHU de Rouen, Hôpital Charles Nicolle, Rouen, Seine Maritime
  - Hôpital Avicenne, Hôpitaux universitaires Paris Seine-, Bobigny, Île-de-France Region
  - Hôpital d'Instruction des Armées Percy, Clamart, Île-de-France Region
  - Hôpital Louis Mourier, Colombes, Île-de-France Region
  - Centre Hospitalier Intercommunal de Créteil, Créteil, Île-de-France Region
  - Centre Hospitalier de Versailles André Mignot, Le Chesnay, Île-de-France Region
  - Hôpital Bicêtre, Le Kremlin-Bicêtre, Île-de-France Region
  - Institut Curie, Paris, Île-de-France Region
  - Hôpital Pitié Salpétrière, Paris, Île-de-France Region
  - Centre Hospitalier Paris Saint-Joseph, Paris, Île-de-France Region
  - Institut Mutualiste Montsouris, Paris, Île-de-France Region
  - Hôpital Européen Georges Pompidou, Paris, Île-de-France Region
  - Hôpital Bichat Claude Bernard, Paris, Île-de-France Region
  - Hôpital Tenon, Paris, Île-de-France Region
  - Centre cardiologique du Nord, Saint-Denis, Île-de-France Region
  - Hôpital Foch, Suresnes, Île-de-France Region
  - Gustave Roussy, Villejuif, Île-de-France Region

IPD SHARING:
Plan to Share IPD: Undecided